CLINICAL TRIAL: NCT05028543
Title: Total Laparoscopic Hysterectomy(TLH) With Prior Uterine Artery Clipping Versus Conventional Total Laparoscopic Hysterectomy
Brief Title: TLH With Prior Uterine Artery Clipping at Its Origin Versus Conventional TLH
Acronym: TLH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Yasmeen Ahmed Mohamed Mohamed Taha, The principal investigator, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: New TLH technique
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Total Laparoscopic Hysterectomy
Keywords: New technique for TLH; Clipping of uterine artery at its origin; Hystrectomy

STUDY DESIGN:
Intervention Model Description: A Randomized controlled Trial.
Who Masked: Investigator
Masking Description: The study design precluded neither participants nor the surgeons will be blinded, only data analyzer will be blinded to each allocation group" single blinded study". However, the outcomes of the study are objective not subjective and will not be affected by lack of blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional TLH (Placebo Comparator): women that will be subjected to conventional Total laparoscopic hysterectomy
  Interventions: Procedure: Conventional TLH
- TLH with prior uterine artery clipping at its origin (Experimental): women that will be subjected to TLH with prior uterine artery clipping at its origin
  Interventions: Procedure: Clipping of utrine artery at its origin before bginning of TLH

INTERVENTIONS:
Procedure: Conventional TLH — Procedure: conventional Total laparoscopic hysterectomy the uterine artery will be identified close to the isthmus then coagulated at this level, close to the uterus , using bipolar diathermy. The utero-vesical fold will be dissected and the bladder will be pushed down done.. The vasculature of the uterus will now secured and this will be evidenced by the pale color of the fundus.
  Using either bipolar diathermy , the cornual pedicles on one side will be desiccated and cut. Also, both the uterosacral and cardinal ligaments will be coagulated and cut. So that, the opposite side pedicles can be taken care of.. The infundibulopelvic ligaments will be coagulatd and cut if it is necessary to remove both ovaries. A vaginal cuff was inserted into the vagina to identify the vault, which will then cut laparoscopically using a monopolar hook, where the specimen will be completely detached.
  Arms: conventional TLH
Procedure: Clipping of utrine artery at its origin before bginning of TLH — the uterine artery will be dissected using posteriorly and medially to the infundibulopelvic ligament, the ureter should be first identified. The surgeon may grab the obliterated umbilical artery at the anterior abdominal wall and retract it. The movement of the umbilical artery may be Seen at the ovarian fossa perpendicular to the ureter
  The uterine vessels will be clipped at their origin from the hypogastric vessels using aclip applier which will be introduced through 10mm trocar. clipping of the artery will be performed through application of two 5 mm size metallic clips in continuity and complete the laparoscopic hysterectomy with the same steps of the conventional method.
  Arms: TLH with prior uterine artery clipping at its origin

SUMMARY:
A randomized controlled trial was done on 30 women planned for TLH, and divided into two groups; group A includes women that will be subjected to conventional TLH, and group B includes women that will be subjected to TLH with prior uterine artery clipping at its origin. Both grouped will be compared regarding the blood loss, operation time, intraoperative complications and post-operative follow-up

DETAILED DESCRIPTION:
Patients will be randomized into 2 groups:

Group (A): Women who will be subjected to conventional Total laparoscopic hysterectomy Group (B): Women who will be subjected to Total laparoscopic hysterectomy with prior uterine artery clipping at its origin.

Intraoperative:

Pre-Anesthesia medications: All patients will receive intravenous antibiotics 30 minutes before induction of anesthesia {Cefotaxime 1gm (Claforan®-EIPICO) & Metronidazole 500 mg (Flagyl®-rPr)}.

* All patients will be positioned in the dorsal lithotomy position
* Examination under anesthesia will be done to assess uterine size, mobility and the presence of any gross adnexal pathology.
* A bladder catheter will be placed to empty the bladder and to monitor the urine output.
* A uterine manipulator (V care cup®) will be placed through the cervix to manipulate the uterus.
* The surgeon will stay on the left side of the patient, the assistant on the right side and the scrub nurse in between the patient's legs for uterine manipulation.
* A small vertical incision will be made into the depth of the supra umbilicus about 0.5 cm length;
* The closed method will be employed where the Veress needle will be inserted vertically into the supra -umbilical incision.
* Hanging drop test will be done to ensure proper needle placement through attaching an open syringe filled with saline to the Veress needle and observing the drop.
* Insertion of 10 mm trocar through the supra umbilical incision and then the operating laparoscope will be inserted through the supra umbilical port.
* CO2 Insufflation will be started to induce pneumoperitoneum till pressure reached 20 mmHg and reduced to 15 mm afterwards.
* Two 5 mm lower quadrant ancillary trocars will be inserted lateral to the inferior epigastric arteries under direct laparoscopic vision above the pubic hairline.
* Another 10 mm trocar will be inserted 3cm above the left lower ancillary trocar under direct vision.

Technical aspects After a thoroughly exploration of the pelvic cavity, the entire abdomen will be surveyed before starting the procedure.

The size of the uterus, presence of myomas, and adnexa and course of ureters will be visualized.

1. In conventional TLH (control group) :The following will be done 1. -Round ligaments will be coagulated and cut. 2. -Separation of the adnexal structures from the uterine corpus for subsequent preservation or removal:

   1. For salpingo-oophorectomy: the infundibulopelvic ligament will be placed on contralateral traction, awindow will be created in the medial leaf of the broad ligament below the ovarian vessels and ventral to the ureter, maintaining direct visualization of the

      ureter.The infundibulopelvic ligament will be coagulated and divided.
   2. If preservation of the adnexa will be planned:The fallopian tube and utero-ovarian ligament will be coagulated close to the uterine fundus and detached. The medial leaf of the broad ligament can be incised down to a level just ventral to the pelvic ureter to allow the adnexa to drop out of the field of dissection. The procedure will be repeated on the contralateral side 3. -Dissecting, occluding, and dividing the blood supply prior to extirpation of the uterine corpus:(skeletonization of the uterine vessels at uterine isthmus, coagulation of the vessels, after identification of the ureter) 4. Transection of the cardinal ligament complex with colpotomy and amputation of the cervix from the vaginal apex.

      5. Removing the specimen. 6. Laparoscopic closure of the vaginal cuff.
2. In intervention group:

The same steps as in control group but with extra step after coagulation and cutting of the round ligaments. The following steps will be done to reach to the origin of uterine artery from internal iliac artery :

Posterior and medial to the infundibulopelvic ligament, the ureter should be first identified. The surgeon may grab the obliterated umbilical artery at the anterior abdominal wall and retract it. The movement of the umbilical artery may be Seen at the ovarian fossa perpendicular to the ureter.

The peritoneum of the ovarian fossa should be opened above the ureter and over the impression of the umbilical artery. The ureter will be retracted medially and the umbilical artery will be dissected vertical and cranially. Usually, one will identify the origin of the uterine artery at this point, which goes medial to the umbilical artery and almost parallel to the ureter. The uterine vessels will be clipped at their origin from the hypogastric vessels using aclip applier which will be introduced through 10mm trocar. clipping of the artery will be performed through application of two 5 mm size metallic clips in continuity and complete the laparoscopic hysterectomy with the same steps of the conventional method

Postoperative care:

1. The patient will receive IV fluids in the first 24hours (3litres).
2. Oral clear fluid intake will be started 8 hours after the operation.
3. Another dose of antibiotics will be received 6hrs after the operation with the same regimen used in induction.
4. Postoperative analgesia (NSIDS ®)
5. The urinary catheter will be removed after 24hrs after the operation.
6. CBC will be withdrawn 24hrs after the operation.
7. Histopathological examination of the specimen will be done.
8. Vaginal douches and coital activity will be advised against for 3 monthes

ELIGIBILITY:
Inclusion Criteria:

* • Benign conditions as indications for hysterectomy (e.g., dysfunctional uterine bleeding, adenomyosis and uterine fibroids) provided that the uterus size is no more than 14 weeks.

Exclusion Criteria:

* • Obese patients i.e., BMI > 35 k.g\m2.

  * Suspected extensive pelvic adhesions based on previous history and examination.
  * Factors which may delay vaginal vault healing as uncontrolled diabetes, prolonged corticosteroid therapy or advanced liver diseases.
  * Inability to give adequate informed consent to participate in the study.
  * Previous ureteric surgery
  * Previous midline incision
  * Previous uterine artery embolization.
  * Known tubo ovarian pathology requiring primary laparotomy, e.g. large adnexal masses.
  * Conditions interfering with laparoscopic surgery e.g. significant cardiopulmonary disease.
  * Large uterus interfering with TLH (size >14 gestational weeks).
  * Broad ligament and cervical myoma hindering access to the lateral pelvic wall
  * Having endometriosis grade III orIV according to ASRM classification.
  * . Having 2nd or 3rd degree uterine descent

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2021-08-21 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-08-21 (Estimated)

PRIMARY OUTCOMES:
The total blood loss | start time is the insertion of 10 mm telescope trocar end-time is the removal of all trocars
  Blood loss (mL): The total blood loss will be from the suction apparatus

SECONDARY OUTCOMES:
intraoperative or postoperative complications | during the Laparoscopy and during the hospital stay (24 hours postoperative
  intraoperative complications are that during the Laparoscopy postoperative complications are that during the hospital stay (24 hours postoperative)

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Elgndi, MD, Study Director — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gueli Alletti S, Restaino S, Finelli A, Ronsini C, Lucidi A, Scambia G, Fanfani F. Step by Step Total Laparoscopic Hysterectomy with Uterine Arteries Ligation at the Origin. J Minim Invasive Gynecol. 2020 Jan;27(1):22-23. doi: 10.1016/j.jmig.2019.06.001. Epub 2019 Jun 12. PMID 31201941
- [Background] BriJtow R:Total Laparoscopic Hystrectomy: Text book of Te Linde's Atlas Operative Gynecology Robert E, Bristow Ricardo Azziz Robert E.Bristo. 10thEdition. (2014b); ch.4: 35-41
- [Background] DOS SANTOS MARTIN, R. L.,et al: How do I perform temporary occlusion of the uterine arteries during laparoscopic myomectomy. Gynecol Obstet (Sunnyvale), 2015, 5.278: 2161-0932.1000278.
- [Background] Johanson ML, Lieng M. Changes in route of hysterectomy in Norway since introduction of robotic approach. Facts Views Vis Obgyn. 2021 Mar 31;13(1):35-40. doi: 10.52054/FVVO.13.1.005. PMID 33889859
- [Background] Kale A, Aksu S, Terzi H, Demirayak G, Turkay U, Sendag F. Uterine artery ligation at the beginning of total laparoscopic hysterectomy reduces total blood loss and operation duration. J Obstet Gynaecol. 2015;35(6):612-5. doi: 10.3109/01443615.2014.990431. Epub 2014 Dec 17. PMID 25517762
- [Background] Popa A, Copaescu C, Horhoianu V. Laparoscopic total hysterectomy still not routinely chosen Operative description and available instruments. J Med Life. 2019 Jul-Sep;12(3):301-307. doi: 10.25122/jml-2019-0051. PMID 31666835
- [Background] Howard W Jones III MD and J. A. R. M:Te Linde's Operative Gynecology ( 11th Edition) 2015
- [Background] Zhao D, Li B, Wang Y, and Liu S, Zhang Yand Zhang G: